CLINICAL TRIAL: NCT02624661
Title: Glycerol Block of the Trigeminal Ganglion in Trigeminal Neuralgia Using a New Neuronavigation-based Surgical Technique
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: technical problems
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/1192
Record Dates: First submitted 2015-11-26; First posted 2015-12-08 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Trigeminal Neuralgia; Headache Disorders
Keywords: Trigeminal ganglion; Glycerol; Nerve block
MeSH Terms: conditions — Trigeminal Neuralgia; Headache Disorders | interventions — Glycerol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glycerol injection (Experimental): The patients will be injected with glycerol using a new neuronavigation-based technique in the trigeminal ganglion.
  Interventions: Drug: Glycerol

INTERVENTIONS:
Drug: Glycerol

SUMMARY:
Trigeminal neuralgia is one of the strongest pains known to humans. Some patients do not have enough effect with the available pharmaceutical treatments and are offered a type of surgery, which involves the injection of glycerol in a nerve structure called trigeminal ganglion. The researchers will do a pilot study on 10 patients with a new surgical technique using neuronavigation. The researchers believe that this new neuronavigation-based system can improve the precision of the technique and reduce the risk for complications.

ELIGIBILITY:
Inclusion Criteria:

* Informed and written consent
* Trigeminal neuralgia defined in International Classification of Headache Disorders (ICHD)-3 criteria
* Unsatisfactory effect of pharmacological treatment

Exclusion Criteria:

* Microvascular decompression is seen as a better alternative
* Heart or lung disease
* Any kind of systematic or local disease or illness that may significantly increase the risk of complications for the procedure related to injection
* Psychiatric illness that hinders participation in the study
* Known pregnancy or breast feeding
* Inadequate use of contraceptives
* Overuse or abuse of opioids
* Abuse of medications, narcotics or alcohol
* Anomalies which hinder or impede the used method of injection
* Allergy or any other hypersensitivity reactions against marcain, lidocaine, xylocain or adrenalin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | For the follow-up period of 12 weeks
  Number of adverse events and number of participants with adverse events after glycerol injection in the trigeminal ganglion and severity of adverse events by the method used. Registration of any adverse events categorized by probable relationship to drug or the procedure. Data obtained from the headache diaries as well as open questions during consultations.

SECONDARY OUTCOMES:
Number of attacks with trigeminal neuralgia | 12 weeks
Intensity of the trigeminal neuralgia attacks assessed by Visual analogue scale | 12 weeks
  expressed as score on Visual analogue scale (VAS) for pain
Intensity of the trigeminal neuralgia attacks assessed by questionnaire | 12 weeks
  expressed by means of patient global impression of change questionnaire (PGIC)
Number of doses of common analgesics | 12 weeks
  week 1-4, week 5-8, week 9-12

CONTACTS AND LOCATIONS:
Overall Officials: Erling A Tronvik, PhD, MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of Neuroscience, Norwegian University of Science and Technology, Trondheim, Norway